CLINICAL TRIAL: NCT06065748
Title: A Phase III Randomized, Open-Label Study Evaluating Efficacy and Safety of Giredestrant Compared With Fulvestrant, Both Combined With a CDK4/6 Inhibitor, in Patients With Estrogen Receptor-Positive, HER2-Negative Advanced Breast Cancer With Resistance to Prior Adjuvant Endocrine Therapy
Brief Title: A Study to Evaluate Efficacy and Safety of Giredestrant Compared With Fulvestrant (Plus a CDK4/6 Inhibitor), in Participants With ER-Positive, HER2-Negative Advanced Breast Cancer Resistant to Adjuvant Endocrine Therapy (pionERA Breast Cancer)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO44657; 2022-502980-39-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Estrogen Receptor-Positive, HER2-Negative Advanced Breast Cancer
Keywords: oral Selective Estrogen Receptor Degrader (SERD); CDK4/6 inhibitor (CDK4/6i); ESR1 mutation
MeSH Terms: interventions — giredestrant; Fulvestrant; abemaciclib; palbociclib; ribociclib; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Giredestrant + Investigator's Choice of CDK4/6i (Experimental): Participants in the experimental arm will receive giredestrant plus the investigator's choice of CDK4/6 inhibitor (CDK4/6i): palbociclib, ribociclib, or abemaciclib.
  Interventions: Drug: Giredestrant; Drug: Abemaciclib; Drug: Palbociclib; Drug: Ribociclib; Drug: LHRH Agonist; Diagnostic Test: FoundationOne Liquid CDx Assay (F1LCDx)
- Fulvestrant + Investigator's Choice of CDK4/6i (Active Comparator): Participants in the control arm will receive fulvestrant plus the investigator's choice of CDK4/6 inhibitor (CDK4/6i): palbociclib, ribociclib, or abemaciclib.
  Interventions: Drug: Fulvestrant; Drug: Abemaciclib; Drug: Palbociclib; Drug: Ribociclib; Drug: LHRH Agonist; Diagnostic Test: FoundationOne Liquid CDx Assay (F1LCDx)

INTERVENTIONS:
Drug: Giredestrant — Giredestrant 30 milligrams (mg) orally (PO) once a day (QD) on Days 1-28 of each 28-day cycle until progressive disease (PD) or unacceptable toxicity.
  Other Names: RO7197597; RG6171; GDC-9545
  Arms: Giredestrant + Investigator's Choice of CDK4/6i
Drug: Fulvestrant — Fulvestrant 500 mg intramuscularly (IM) on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent 28-day cycle until PD or unacceptable toxicity.
  Arms: Fulvestrant + Investigator's Choice of CDK4/6i
Drug: Abemaciclib — If chosen by the investigator as the CDK4/6i, participants will receive abemaciclib 150 mg PO twice per day (BID) on Days 1-28 of each 28-day cycle until PD or unacceptable toxicity.
Drug: Palbociclib — If chosen by the investigator as the CDK4/6i, participants will receive palbociclib 125 mg PO QD on Days 1-21 of each 28-day cycle until PD or unacceptable toxicity.
Drug: Ribociclib — If chosen by the investigator as the CDK4/6i, participants will receive ribociclib 600 mg PO QD on Days 1-21 of each 28-day cycle until PD or unacceptable toxicity.
Drug: LHRH Agonist — Only pre/perimenopausal female participants and male participants will receive a luteinizing hormone-releasing hormone (LHRH) agonist locally approved for use in breast cancer on Day 1 of each 28-day treatment cycle.
Diagnostic Test: FoundationOne Liquid CDx Assay (F1LCDx) — F1LCDx is a next-generation sequencing (NGS)-based in vitro diagnostic test that detects and analyses genomic alterations in circulating cell-free DNA (cfDNA) isolated from plasma derived from the anti-coagulated peripheral whole blood of cancer patients. It will be used to determine the eligibility of participants requiring confirmation of ESR1 mutation status (mutation detected [ESR1m] vs. no mutation detected [ESR1nmd]).
  Other Names: F1LCDx

SUMMARY:
This is a Phase III, randomized, open-label multicenter study that will evaluate the efficacy and safety of giredestrant compared with fulvestrant, both in combination with the investigator's choice of a CDK4/6 inhibitor (palbociclib, ribociclib or abemaciclib), in participants with estrogen receptor-positive (ER+), human epidermal growth factor receptor 2-negative (HER2-) advanced breast cancer who have developed resistance to adjuvant endocrine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic adenocarcinoma of the breast, not amenable to treatment with curative intent
* Documented estrogen receptor-positive (ER+), HER2-negative (HER2-) tumor assessed locally on the most recent tumor biopsy (or an archived tumor sample if a recent tumor sample is not available for testing)
* Confirmed ESR1 mutation status (ESR1m versus ESR1nmd) in baseline circulating tumor DNA (ctDNA) through central laboratory testing
* Resistance to prior adjuvant endocrine therapy (ET), which is defined as having relapsed with prior standard adjuvant ET, on-treatment after >/=12 months or off-treatment within 12 months of completion. Prior use of adjuvant CDK4/6i is allowed (if relapse occurred >/=12 months since completion).
* No prior systemic anti-cancer therapy for advanced disease
* Measurable disease as defined per RECIST v.1.1 or non-measurable (including bone-only) disease
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1
* For pre/perimenopausal women and for men: willing to undergo and maintain treatment with approved LHRH agonist therapy (as per local guidelines) for the duration of study treatment

Exclusion Criteria:

* Prior systemic therapy (e.g., prior chemotherapy, immunotherapy, or biologic therapy) for locally advanced unresectable or metastatic breast cancer
* Prior treatment with another SERD (e.g., fulvestrant, oral SERDs) or novel ER-targeting agents
* Advanced, symptomatic, visceral spread that is at risk of life-threatening complications in the short term
* Active cardiac disease or history of cardiac dysfunction
* Clinically significant history of liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2023-12-11 (Actual); Primary Completion 2027-02-19 (Estimated); Study Completion 2029-02-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) in the ESR1 mutation (ESR1m) Subgroup | From randomization to first occurrence of progressive disease (PD) or death (up to 5 years)
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), or death from any cause during the study.
PFS in the Full Analysis Set (FAS) Population | From randomization to first occurrence of PD or death (up to 5 years)

SECONDARY OUTCOMES:
PFS in the ESR1 no-mutation-detected (ESR1nmd) Subgroup | From randomization to first occurrence of PD or death (up to 5 years)
Overall Survival (OS) | From randomization until death from any cause (up to 5 years)
  OS is defined as the time from randomization to death from any cause. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Confirmed Objective Response Rate (cORR) | From randomization until treatment discontinuation (up to 5 years)
  The cORR is defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions at least 4 weeks apart, as determined by the investigator according to RECIST v1.1. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Duration of Response (DOR) | From the first occurrence of a documented objective response to PD or death (up to 5 years)
  DOR is defined as the time from the first occurrence of a documented objective response to PD, as determined by the investigator according to RECIST v1.1, or death from any cause (whichever occurs first). It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Clinical Benefit Rate (CBR) | From randomization until treatment discontinuation (up to 5 years)
  The CBR is defined as the percentage of participants with stable disease for at least (≥)24 weeks or a CR or PR, as determined by the investigator according to RECIST v1.1. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Time to Chemotherapy | From randomization until the start of chemotherapy or death (up to 5 years)
  Time to chemotherapy is defined as the time from randomization until the start date of the first chemotherapy or death from any cause (whichever occurs first). It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Time to Confirmed Deterioration (TTCD) in Pain Severity | From randomization until end of follow-up (up to 5 years)
  TTCD in pain severity is defined as the time from randomization to the first documentation of ≥2-point increase from baseline on the "worst pain" item score of the Brief Pain Inventory-Short Form (BPI-SF). It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
TTCD in Pain Presence and Interference | From randomization until end of follow-up (up to 5 years)
  TTCD in pain presence and interference is defined as the time from randomization to the first documentation of ≥10-point increase in pain score, as determined using the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 (EORTC QLQ-C30) questionnaire. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
TTCD in Physical Functioning | From randomization until end of follow-up (up to 5 years)
  TTCD in physical functioning (PF) is defined as the time from randomization to the first documentation of ≥10-point decrease in PF score, as determined using the EORTC QLQ-C30 questionnaire. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
TTCD in Role Functioning | From randomization until end of follow-up (up to 5 years)
  TTCD in role functioning (RF) is defined as the time from randomization to the first documentation of ≥10-point decrease in RF score, as determined using the EORTC QLQ-C30 questionnaire. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
TTCD in Global Health Status/Quality of Life | From randomization until end of follow-up (up to 5 years)
  TTCD in in Global Health Status/Quality of Life (GHS/QoL) is defined as the time from randomization to the first documentation of ≥10-point decrease in GHS/QoL score, as determined using the EORTC QLQ-C30 questionnaire. It will be analyzed in the FAS and in the ESR1m and ESR1nmd subgroups.
Incidence and Severity of Adverse Events | From Baseline until 28 days after the final dose of study treatment (up to 5 years)
  Incidence will be reported as the number of participants with at least one adverse event, with severity determined according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5 (NCI CTCAE v5.0).
Number of Participants with Vital Sign Abnormalities Over the Course of the Study | From Baseline until 28 days after the final dose of study treatment (up to 5 years)
  Vital signs include respiratory rate, pulse rate, systolic and diastolic blood pressure, and temperature.
Number of Participants with Clinical Laboratory Test Abnormalities for Hematology and Biochemistry Parameters Over the Course of the Study | From Baseline until 28 days after the final dose of study treatment (up to 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (351):
- United States (61):
  - Southern Cancer Center, Daphne, Alabama
  - Sutter Auburn Faith Hospital, Auburn, California
  - La Hematology Oncology Medical Group, Glendale, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Cancer Center, Newport Beach, California
  - Sutter Medical Group, Roseville Clinic, Roseville, California
  - Sutter Health Medical Center, Sacramento, California
  - The Lundquist Institute for BioMedical Innovation at Harbor-UCLA Medical Cente, Torrance, California
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - MedStar Washington Hosp Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - Florida Cancer Specialists - Broadway, Fort Myers, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Florida Cancer Specialists - Tampa, Tampa, Florida
  - Florida Cancer Specialists - EAST - SCRI - PPDS, West Palm Beach, Florida
  - Grady Health System, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Mission Cancer + Blood - IMMC, Des Moines, Iowa
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Hamburg, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Maryland Oncology Hematology, Annapolis, Maryland
  - Frederick Health Hospital, Frederick, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - HCA Midwest Division, Kansas City, Missouri
  - Cancer Care Center of O'Fallon, O'Fallon, Missouri
  - Oncology Hematology West - Grand Island, Grand Island, Nebraska
  - Oncology Hematology West - Legacy, Omaha, Nebraska
  - Astera Cancer Care East Brunswick, East Brunswick, New Jersey
  - Capital Health Regional Medical Center, Pennington, New Jersey
  - Queens Hospital Cancer Center, Jamaica, New York
  - Duke Women Cancer Care, Raleigh, North Carolina
  - Oncology Hematology Care, Cincinnati, Ohio
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Alliance Cancer Specialists, Bensalem, Pennsylvania
  - Ann B. Barshinger Cancer Institute, Lancaster, Pennsylvania
  - Abramson Cancer Center; Univ of Pennsylvania; Clinical Research Unit, Philadelphia, Pennsylvania
  - WellSpan Oncology Research, York, Pennsylvania
  - Brown University Health, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute - Aberdeen, Aberdeen, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - West Cancer Center, Germantown, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology Cancer Center, Austin, Texas
  - JPS Oncology & Infusion Center, Fort Worth, Texas
  - Texas Oncology - DFW, Irving, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
  - West Virginia University Hospitals Inc, Morgantown, West Virginia
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora St Lukes Medical Center, Milwaukee, Wisconsin
- Argentina (10):
  - Centro de Investigaciones Médicas y Desarrollo LC S.R.L, Buenos Aires
  - Inst. de Oncologia Angel H. Roffo, Buenos Aires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
  - Sanatorio Allende, Córdoba
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Hospital Alemán, Recoleta
  - Instituto de Oncología de Rosario, Rosario
  - Sanatorio Parque S.A., Rosario
  - Hospital Provincial del Centenario, Rosario
  - Centro Oncológico de Excelencia, San Juan
- Australia (9):
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Mater Hospital, North Sydney, New South Wales
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Mater Misericordiae Limited, South Brisbane, Queensland
  - Cancer Research SA, Adelaide, South Australia
  - Barwon Health, Geelong, Victoria
  - Sunshine Hospital, St Albans, Victoria
  - South West Healthcare, Warrnambool, Victoria
- Austria (5):
  - Lkh-Univ. Klinikum Graz, Graz
  - Medical University Innsbruck, Innsbruck
  - Ordensklinikum Linz Barmherzige Schwestern, Linz
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
  - Medizinische Universität Wien, Vienna
- Belgium (8):
  - Cliniques Universitaires St-Luc, Brussels
  - GHdC Site Les Viviers, Charleroi
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège (Sart Tilman), Liège
  - AZ St Maarten Campus Leopoldstr, Mechelen
  - Clinique Ste-Elisabeth, Namur
  - ZAS Sint Augustinus Wilrijk, Wilrijk
- Brazil (20):
  - Crio - Centro Regional Integrado de Oncologia, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Obras Sociais Irma Dulce - Osid, Salvador, Estado de Bahia
  - Hospital Sírio-Libanês, Brasília, Federal District
  - Hospital Araujo Jorge, Goiânia, Goiás
  - Hospital Sao Domingos, São Luís, Maranhão
  - Hospital do Câncer de Londrina, Londrina, Paraná
  - Hospital do Cancer de Pernambuco - HCP, Recife, Pernambuco
  - Vencer Oncoclínica - Centro de Pesquisa do Piauí, Teresina, Piauí
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Hospital A. C. Camargo, São Paulo, São Paulo
  - Instituto D'Or de Pesquisa e Ensino, Rio de Janeiro
- Canada (16):
  - Cross Cancer Institute, Edmonton, Alberta
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Credit Valley Hospital/Carlo Fidani Peel Regional Cancer Centre, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
  - North York General Hospital, Toronto, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - CIUSSS du Saguenay Lac-Saint-Jean, Chicoutimi Hospital, Chicoutimi, Quebec
  - CISSS Chaudière-Appalaches, Lévis, Quebec
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - CHU de Québec - Hôpital du Saint-Sacrement, Québec, Quebec
  - Hopital regional de saint jerome, Saint-Jérôme, Quebec
  - Centre hospitalier regional de Trois-Rivieres, Trois-Rivières, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Chile (7):
  - Hospital las Higueras, Concepción, Región Bio Bio
  - Centro de Oncología de Precisión, Las Condes
  - Clínica Puerto Montt, Port Montt
  - Oncovida, Providencia
  - Centro De Cancer Universidad Catolica, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Icegclinic, Santiago
- China (29):
  - Beijing Cancer Hospital, Beijing
  - the First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital, Chongqing Medical University, Chongqing
  - Fujian Medical University Union Hospital, Fuzhou
  - No. 900 Hospital (Fuzhou General Hospital), Fuzhou
  - Cancer Center, Sun Yat-sen University of Medical Sciences, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jinan Central Hospital, Jinan
  - Shandong Cancer Hospital, Jinan
  - The First People's Hospital of Yunnan Province, Kunming
  - The First Affiliated Hospital to Henan University of Science and Technology, Luoyang
  - Guangxi Cancer Hospital of Guangxi Medical University, Nanning
  - Zhongshan Hospital Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanxi Province Cancer Hospital, Taiyuan
  - Taizhou Hospital of Zhejiang Province, Taizhou
  - Tianjin Cancer Hospital, Tianjin
  - The Tumor Hospital of Xinjiang Medical University, Ürümqi
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiao Tong University, Xi'an
  - Xi'an International Medical Center Hospital, Xi'an
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Zhejiang Cancer Hospital, Zhejiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
- Colombia (5):
  - Fundación CTIC - Centro de Tratamiento e Investigación sobre Cáncer Luis Carlos Sarmiento Angulo, Bogota, D.C.
  - Clinica Colsanitas S.A. sede Clinica Universitaria Colombia, Bogotá D.C.
  - IPS Salud SURA Chipichape Cali, Cali
  - Oncomedica S.A., Montería
  - Sociedad de Oncología y hematología del Cesar Ltda, Valledupar
- Costa Rica (3):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
  - Proclinical Pharma, San José
- Finland (2):
  - Kuopio Uni Hospital, Kuopio
  - Tampere University Hospital, Tampere
- France (13):
  - ICO Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz, Besançon
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Saint Louis, La Rochelle
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Cancerologie Grand Montpellier, Montpellier
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - IUCT Oncopole, Toulouse
  - Gustave Roussy, Villejuif
- Germany (11):
  - Sozialstiftung Bamberg, Klinikum am Bruderwald, Gynäkologie, Bamberg
  - St. Elisabeth Krankenhaus Köln GmbH, Cologne
  - DONAU ISAR Klinikum Deggendorf, Deggendorf
  - Gynonco Düsseldorf, MVZ Medical Center GmbH, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Essen
  - Praxis für Interdisziplinäre Onkologie und Hämatologie GbR, Freiburg im Breisgau
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Brustzentrum Rhein-Ruhr Servicegesellschaft mbH, Mönchengladbach
  - Rotkreuzklinikum München, München
- Greece (5):
  - Anticancer Hospital Ag. Savas, Athens
  - Aretaieio Hospital of Athens, Athens
  - University Hospital of Larissa, Larissa
  - University Hospital of Patras Medical Oncology, Pátrai
  - European Interbalkan Medical Center, Thessaloniki
- Guatemala (7):
  - Oncomedica, Guatemala City
  - Celan S.A., Guatemala City
  - INTEGRA Cancer Institute, Guatemala City
  - Onco Go, S.A., Guatemala City
  - Grupo Angeles, Guatemala City
  - Medi-k, Guatemala City
  - Centro Medico Integral de Cancerologia CEMIC, Salcajá
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Bács-Kiskun Vármegyei Oktatókórház, Kecskemét
  - B-A-Z Vármegyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
  - Nograd Varmegyei Szent Lazar Korhaz, Salgótarján
- India (8):
  - HealthCare Global Enterprises Limited, Banglore, Karnataka
  - MVR Cancer Centre and Research Institute, Kozhikode, Kerala
  - Regional Cancer Centre, Trivandrum, Kerala
  - Sir H. N. Reliance Foundation Hospital and Research Centre, Mumbai, Maharashtra
  - Grant Medical Foundation, Ruby Hall Clinic, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Sunact Cancer Institute, Thane, Maharashtra
  - Max Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
- Israel (4):
  - Hadassah Ein Karem Hospital, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba MC, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (21):
  - Presidio Ospedaliero di Summa-Perrino, Brindisi, Apulia
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialita San Giuseppe Moscati, Avellino, Campania
  - Azienda Ospedaliera Universitaria Federico II, Napoli, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - I.R.S.T Srl IRCCS, Meldola, Emilia-Romagna
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - RCCS - Centro di Riferimento, Aviano (PN), Friuli Venezia Giulia
  - A.O. Universitaria S. Maria Della Misericordia Di Udine, Udine, Friuli Venezia Giulia
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - Università Campus Bio-Medico di Roma, Rome, Lazio
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Asst Di Cremona, Cremona, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
  - Humanitas Centro Catanese Di Oncologia, Misterbianco (CT), Sicily
  - Ospedale Di Macerata, Macerata, The Marches
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
- University of Nairobi - Institute of Tropical and Infectious Diseases, Nairobi, Kenya
- Mexico (9):
  - Panamerican Clinical Research S.A de C.V., Guadalajara, Jalisco
  - RENATI INNOVATION S.A.P.I. de C.V, Guadalajara, Jalisco
  - Productos y Servicios Oncologicos Acacias SA de CV, Mexico City, Mexico CITY (federal District)
  - Centro de Atencion Oncologica Viva S de RL de CV, Mexico City, Mexico CITY (federal District)
  - Hospital Zambrano Hellion TecSalud, Monterrey, Nuevo León
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City, Oaxaca
  - PanAmerican Clinical Research, Querétaro, Queréaro, Querétaro
  - CENEIT Oncologicos, Mexico City
  - Clinica Alivia sucursal Coyoacan, Mexico City
- New Zealand (3):
  - Christchurch Hospital, Christchurch
  - Palmerston North Hospital, Palmerston North
  - Whangarei Hospital, Whangarei
- Peru (11):
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital Goyeneche, Arequipa
  - Clínica Santa Beatriz, Lima
  - Hospital Nacional Arzobispo Loayza, Lima
  - Oncosalud Sac, Lima
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica Internacional, Sede San Borja, Lima
  - Instituto Peruano de Oncología y Radioterapia, Lima
  - Clinica San Antonio;Investigaciones Trujillo S.A.C., Trujillo
  - Clinica Peruana Americana, Trujillo
  - Instituto Regional de Enfermedades Neoplasicas - IREN Norte, Trujillo
- Poland (12):
  - Instytut "Centrum Zdrowia Matki Polki", ?ód?
  - Centrum Onkologii im. Prof. Franciszka ?ukaszczyka, Bydgoszcz
  - Szpital Morski Im. Pck, Gdynia
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - ?wi?tokrzyskie Centrum Onkologii, Kielce
  - Przychodnia Lekarska KOMED, Roman Karaszewski, Konin
  - Szpital Wojewódzki im. Miko?aja Kopernika, Koszalin
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli, Lublin
  - Opolskie Centrum Onkologii, Opole
  - Mazowiecki Szpital Wojewódzki im. ?w. Jana Paw?a II, Siedlce
  - Zachodniopomorskie Centrum Onkologii, Szczecin
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
- Portugal (5):
  - IPO de Coimbra, Coimbra
  - Hospital de S. Francisco Xavier, Lisbon
  - Hospital da Luz, Lisbon
  - IPO do Porto, Porto
  - CHVNG/E_Unidade 1, Vila Nova de Gaia
- PanOncology Trials, San Juan, Puerto Rico
- Romania (7):
  - Spitalul Clinic Filantropia, Bucharest
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu, Bucharest
  - Amethyst Cluj, Cluj County
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj Napoca, Cluj-Napoca
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Centrul de Oncologie Oncohelp, Timișoara
- Singapore (3):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
  - Icon Cancer Centre Gleneagles, Singapore
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Africa (3):
  - Cancercare Rondebosch Oncology, Cape Town
  - Cancercare, Port Elizabeth
  - Steve Biko Academic Hospital, Pretoria
- South Korea (10):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hosiptal, Ulsan
- Spain (15):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Virgen de La Arrixaca, EL Palmar (EL Palmar), Murcia
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Dexeus - Grupo Quironsalud, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Juan Ramon Jimenez, Huelva
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico, Jaén
  - Centro Oncologico MD Anderson Internacional, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
- Taiwan (6):
  - Hsin-Chu Branch of National Taiwan University Hospital, Hsinchu
  - China Medical University Hospital, Taichung
  - Veterans General Hospital, Taipei
  - National Taiwan Uni Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Veterans General Hospital - Taichung, Xitun Dist.
- Thailand (6):
  - Chulalongkorn Hospital, Bangkok
  - National Cancer Institute, Bangkok
  - Rajavithi Hospital, Bangkok
  - Chulabhorn Hospital, Lak Si
  - Maharaj Nakorn Chiang Mai Hospital;Depart of Radiology, Muang Chiang MAI Delivery Branch 3
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (8):
  - Sakarya Training and Research Hospital, Adapazarı
  - Ankara City Hospital, Ankara
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Goztepe Prof.Dr. Suleyman Yalcin City Hospital, Kadiköy
  - Mersin City Education and Research Hospital, Mersin
  - Medikal Park Samsun, Samsun
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing